CLINICAL TRIAL: NCT01712399
Title: An Open-label Extension Study to Evaluate the Long-term Safety of Mavrilimumab in Adult Subjects With Rheumatoid Arthritis
Brief Title: A Long Term Safety Study of Mavrilimumab in Adult Subjects With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated after approximately 3 years due to future clinical development plans, including ethical considerations.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-IA-CAM-3001-1109; Earth Explorer X (Other: MedImmune)
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — mavrilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mavrilimumab 100 mg (Experimental): Participants will receive 100 mg mavrilimumab once in every 2 weeks (Q2W) subcutaneously for up to 3 years.
  Interventions: Biological: Mavrilimumab 100 mg

INTERVENTIONS:
Biological: Mavrilimumab 100 mg — Participants will receive 100 mg mavrilimumab once in every 2 weeks (Q2W) subcutaneously for up to 3 years

SUMMARY:
A clinical study to investigate the safety of mavrilimumab, an antibody being developed for the treatment of moderate to severe rheumatoid arthritis, an inflammatory condition that affects the joints.

DETAILED DESCRIPTION:
Despite the therapeutic improvements with recent biologic agents approved for rheumatoid arthritis (RA), there is still a significant unmet medical need for the treatment of subjects with this chronic disease to achieve a faster, more complete response, and higher rates of remission. This study is an open-label extension study for subjects who have participated in one of the qualifying development program studies with mavrilimumab. Participation in this study will allow these subjects to continue to receive long-term treatment with mavrilimumab. The data from this study will provide an evaluation of the long-term safety of mavrilimumab in adult subjects with RA. In addition, long-term exploratory efficacy outcomes such as joint damage and disability will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the treatment period of the qualifying study or will have failed to respond adequately to investigational product at a predefined time point in the qualifying study regardless of their initial randomization.
* No evidence of clinically uncontrolled respiratory disease to be confirmed by a local pulmonologist

Exclusion Criteria:

* Subjects who have been permanently discontinued from investigational product in previous qualifying study.
* Any new conditions or worsening of any pre-existing conditions as defined in the protocol.

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2013-01-28; Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- Argentina (4):
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Ciudad Autonoma de Buenos Aire
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Chile (2):
  - Research Site, Santiago
  - Research Site, Viña del Mar
- Research Site, Barranquilla, Colombia
- Czechia (6):
  - Research Site, Bruntál
  - Research Site, Jihlava
  - Research Site, Ostrava - Trebovice
  - Research Site, Prague
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- Research Site, Tallinn, Estonia
- Germany (2):
  - Research Site, Cologne
  - Research Site, Magdeburg
- Greece (2):
  - Research Site, Athens
  - Research Site, Larissa
- Hungary (4):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
- Israel (3):
  - Research Site, Ashkelon
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
- Research Site, Mérida, Mexico
- Poland (5):
  - Research Site, Gdynia
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Wroclaw
- Russia (5):
  - Research Site, Barnaul
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Niška Banja
- Research Site, Bratislava, Slovakia
- Research Site, Durban, South Africa
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Málaga
  - Research Site, Santiago de Compostela
- Ukraine (5):
  - Research Site, Donetsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Lutsk
  - Research Site, Vinnytsia
- United Kingdom (2):
  - Research Site, Edinburgh
  - Research Site, London

REFERENCES:
- [Derived] Burmester GR, McInnes IB, Kremer JM, Miranda P, Vencovsky J, Godwood A, Albulescu M, Michaels MA, Guo X, Close D, Weinblatt M. Mavrilimumab, a Fully Human Granulocyte-Macrophage Colony-Stimulating Factor Receptor alpha Monoclonal Antibody: Long-Term Safety and Efficacy in Patients With Rheumatoid Arthritis. Arthritis Rheumatol. 2018 May;70(5):679-689. doi: 10.1002/art.40420. Epub 2018 Mar 31. PMID 29361199

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 409 participants consented and 397 participants received mavrilimumab in this study.
Pre-assignment Details: A total of 442 participants who received at least one dose of mavrilimumab provided a pooled analysis of safety and efficacy data from this open-label extension study (CD-IA-CAM-3001-1109) together with the qualifying studies (CD IA CAM 3001 1071 and CD IA CAM 3001 1107).
Groups:
- Mavrilimumab 100 mg: Participants received 100 mg mavrilimumab once in every 2 weeks (Q2W) subcutaneously for up to 3 years.
Period: Overall Study
Arm/Group | Mavrilimumab 100 mg
Started | 397
Completed | 0
Not Completed | 397
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 39
Not completed — Death | 1
Not completed — Adverse Event | 11
Not completed — Study closure | 345

BASELINE CHARACTERISTICS:
Population: The As-treated Population included participants who received at least one dose of mavrilimumab 100 mg every 2 weeks (Q2W).
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339
  Male | 58
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 29
  Asian | 1
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 364
  Other | 2
Region of Enrollment [Number; unit: Participants]
  ARGENTINA | 41
  BULGARIA | 3
  CHILE | 35
  COLOMBIA | 25
  CZECH REPUBLIC | 69
  ESTONIA | 21
  GERMANY | 8
  GREECE | 3
  HUNGARY | 9
  ISRAEL | 11
  MEXICO | 10
  POLAND | 34
  RUSSIAN FEDERATION | 53
  SERBIA | 24
  SLOVAKIA | 1
  SOUTH AFRICA | 2
  SPAIN | 4
  UKRAINE | 39
  UNITED KINGDOM | 5
Weight [Mean (Standard Deviation); unit: Kilogram] | 73.25 (16.40)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received investigational product. A serious adverse event (SAE) was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were defined as AEs with onset date after the first dose of mavrilimumab 100 mg.
Time Frame: From the start of study drug administration up to 12 weeks after the last dose of study drug (approximately up to 3 years)
Population: The As-treated Population included participants who received at least one dose of mavrilimumab 100 mg Q2W.
Measure: Number; unit: Participants
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Participants
  TEAEs | 288
  TESAEs | 46

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Laboratory parameters included hematology, serum chemistry and urinalysis recorded as TEAEs. Clinical laboratory abnormalities recorded as TEAEs were reported.TEAEs were defined as AEs with onset date after the first dose of mavrilimumab 100 mg.
Time Frame: From the start of study drug administration in the study up to 12 weeks after the last dose of study drug (approximately up to 3 years)
Population: The As-treated Population included participants who received at least one dose of mavrilimumab 100 mg Q2W.
Measure: Number; unit: Participants
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Participants
  Anaemia | 8
  Eosinophilia | 1
  Iron deficiency anaemia | 2
  Leukocytosis | 1
  Leukopenia | 1
  Lymphadenopathy | 1
  Neutropenia | 2
  Spontaneous haematoma | 1
  Alanine aminotransferase increased | 8
  Aspartate aminotransferase increased | 6
  Blood creatinine increased | 1
  Blood glucose increased | 1
  Blood pressure increased | 3
  C-reactive protein increased | 1
  Chest X-ray abnormal | 1
  Forced vital capacity abnormal | 1
  Gamma-glutamyltransferase increased | 2
  Hepatic enzyme increased | 2
  Liver function test abnormal | 1
  Mycobacterium tuberculosis complex test positive | 1
  Neutrophil count decreased | 1
  Red blood cell sedimentation rate increased | 1
  Transaminases increased | 3
  Diabetes mellitus | 5
  Dyslipidaemia | 4
  Hypercholesterolaemia | 9
  Hyperglycaemia | 3
  Hyperlipidaemia | 2
  Hypertriglyceridaemia | 2
  Hypoglycaemia | 1
  Type 2 diabetes mellitus | 4

3. Primary Outcome: Number of Participants With Vital Sign Abnormalities Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Vital sign assessments included blood pressure, pulse rate, temperature, weight and respiration rate. Vital sign abnormalities recorded as TEAEs were reported. TEAEs were defined as AEs with onset date after the first dose of mavrilimumab 100 mg.
Time Frame: as for outcome 2
Population: The As-treated Population included participants who received at least one dose of mavrilimumab 100 mg Q2W.
Measure: Number; unit: Participants
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Participants
  Hypertension | 26
  Pyrexia | 3
  Blood pressure increased | 3
  Atrial fibrillation | 1
  Palpitations | 1
  Sinus tachycardia | 1

4. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings Reported as TEAEs
Description: The 12-lead ECG data were summarized and evaluated. TEAEs related to abnormal ECG findings were recorded and reported. TEAEs were defined as AEs with onset date after the first dose of mavrilimumab 100 mg.
Time Frame: as for outcome 2
Population: The As-treated Population included participants who received at least one dose of mavrilimumab 100 mg Q2W.
Measure: Number; unit: Participants
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Participants | 0

5. Primary Outcome: Number of Participants With Forced Expiratory Volume in 1 Second (FEV1) Outside Threshold Values
Description: Pulmonary function testing was performed by spirometry to assess forced expiratory volume in 1 second (FEV1). FEV1 was the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration.The percentage (%) of predicted values of these pulmonary function tests were calculated based on decrease from baseline and categorized as less than or equal to (=<)15% reduction from baseline, greater than (>)15% to =<20% reduction from baseline, >20% reduction from baseline and >20% reduction to <80%. The threshold values refer to baseline values for each participant.
Time Frame: From Week 24 to Week 130 at specified time points
Population: The As-treated Population included participants who received at least one dose of mavrilimumab 100 mg Q2W. Here 'n' represents those participants who were evaluable for this measure at given time points.
Measure: Number; unit: Participants
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Participants
  Week 24:=<15% reduction: number analyzed (Participants) | 236
  Week 24:=<15% reduction | 208
  Week 24:>15% to =<20%: number analyzed (Participants) | 236
  Week 24:>15% to =<20% | 12
  Week 24:>20% reduction: number analyzed (Participants) | 236
  Week 24:>20% reduction | 16
  Week 24:>20% to <80%: number analyzed (Participants) | 236
  Week 24:>20% to <80% | 13
  Week 48:=<15% reduction: number analyzed (Participants) | 231
  Week 48:=<15% reduction | 208
  Week 48: >15% to =<20%: number analyzed (Participants) | 231
  Week 48: >15% to =<20% | 10
  Week 48: >20% reduction: number analyzed (Participants) | 231
  Week 48: >20% reduction | 13
  Week 48:>20% to <80%: number analyzed (Participants) | 231
  Week 48:>20% to <80% | 8
  Week 78:=<15% reduction: number analyzed (Participants) | 178
  Week 78:=<15% reduction | 154
  Week 78:>15% to =<20%: number analyzed (Participants) | 178
  Week 78:>15% to =<20% | 8
  Week 78:>20% reduction: number analyzed (Participants) | 178
  Week 78:>20% reduction | 16
  Week 78:>20% to <80%: number analyzed (Participants) | 178
  Week 78:>20% to <80% | 11
  Week 104:=<15% reduction: number analyzed (Participants) | 29
  Week 104:=<15% reduction | 28
  Week 104:>15% to =<20%: number analyzed (Participants) | 29
  Week 104:>15% to =<20% | 0
  Week 104:>20% reduction: number analyzed (Participants) | 29
  Week 104:>20% reduction | 1
  Week 104:>20% to <80%: number analyzed (Participants) | 29
  Week 104:>20% to <80% | 1
  Week 130:=<15% reduction: number analyzed (Participants) | 3
  Week 130:=<15% reduction | 3
  Week 130:>15% to =<20%: number analyzed (Participants) | 3
  Week 130:>15% to =<20% | 0
  Week 130:>20% reduction: number analyzed (Participants) | 3
  Week 130:>20% reduction | 0
  Week 130:>20% to <80%: number analyzed (Participants) | 3
  Week 130:>20% to <80% | 0

6. Primary Outcome: Number of Participants With Forced Expiratory Volume in 6 Seconds (FEV6) Outside Threshold Values
Description: Pulmonary function testing was performed by spirometry to assess forced expiratory volume in 6 seconds (FEV6). FEV6 was the maximal volume of air exhaled in the six second of a forced expiration from a position of full inspiration. The percentage of predicted values of these pulmonary function tests were calculated based on decrease from baseline and categorized as =<15% reduction from baseline, >15% to =<20% reduction from baseline, >20% reduction from baseline and >20% reduction to <80%. The threshold values refer to baseline values for each participant.
Time Frame: From Week 24 to Week 130 at specified time points
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Participants
  Week 24:=<15% reduction: number analyzed (Participants) | 222
  Week 24:=<15% reduction | 195
  Week 24:>15% to =<20%: number analyzed (Participants) | 222
  Week 24:>15% to =<20% | 14
  Week 24:>20% reduction: number analyzed (Participants) | 222
  Week 24:>20% reduction | 13
  Week 24:>20% to <80%: number analyzed (Participants) | 222
  Week 24:>20% to <80% | 9
  Week 48:=<15% reduction: number analyzed (Participants) | 222
  Week 48:=<15% reduction | 201
  Week 48:>15% to =<20%: number analyzed (Participants) | 222
  Week 48:>15% to =<20% | 13
  Week 48:>20% reduction: number analyzed (Participants) | 222
  Week 48:>20% reduction | 8
  Week 48:>20% to <80%: number analyzed (Participants) | 222
  Week 48:>20% to <80% | 4
  Week 78:=<15% reduction: number analyzed (Participants) | 172
  Week 78:=<15% reduction | 150
  Week 78:>15% to =<20%: number analyzed (Participants) | 172
  Week 78:>15% to =<20% | 8
  Week 78:>20% reduction: number analyzed (Participants) | 172
  Week 78:>20% reduction | 14
  Week 78:>20% to <80%: number analyzed (Participants) | 172
  Week 78:>20% to <80% | 5
  Week 104:=<15% reduction: number analyzed (Participants) | 28
  Week 104:=<15% reduction | 27
  Week 104:>15% to =<20%: number analyzed (Participants) | 28
  Week 104:>15% to =<20% | 0
  Week 104:>20% reduction: number analyzed (Participants) | 28
  Week 104:>20% reduction | 1
  Week 104:>20% to <80%: number analyzed (Participants) | 28
  Week 104:>20% to <80% | 1
  Week 130:=<15% reduction: number analyzed (Participants) | 3
  Week 130:=<15% reduction | 1
  Week 130:>15% to =<20%: number analyzed (Participants) | 3
  Week 130:>15% to =<20% | 0
  Week 130:>20% reduction: number analyzed (Participants) | 3
  Week 130:>20% reduction | 2
  Week 130:>20% to <80%: number analyzed (Participants) | 3
  Week 130:>20% to <80% | 2

7. Primary Outcome: Number of Participants With Forced Vital Capacity (FVC) Outside Threshold Values
Description: Pulmonary function testing was performed by spirometry to assess forced vital capacity (FVC). FVC was the volume of air which can be forcibly exhaled from the lungs after taking the deepest breath possible. The percentage of predicted values of these pulmonary function tests were calculated based on decrease from baseline and categorized as =<15% reduction from baseline, >15% to =<20% reduction from baseline, >20% reduction from baseline and >20% reduction to <80%. The threshold values refer to baseline values for each participant.
Time Frame: From Week 24 to Week 156 at specified time points
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Participants
  Week 24 :=<15% reduction: number analyzed (Participants) | 233
  Week 24 :=<15% reduction | 209
  Week 24:>15% to =<20%: number analyzed (Participants) | 233
  Week 24:>15% to =<20% | 13
  Week 24:>20% reduction: number analyzed (Participants) | 233
  Week 24:>20% reduction | 11
  Week 24:>20% to <80%: number analyzed (Participants) | 233
  Week 24:>20% to <80% | 7
  Week 48:=<15% reduction: number analyzed (Participants) | 239
  Week 48:=<15% reduction | 218
  Week 48:>15% to =<20%: number analyzed (Participants) | 239
  Week 48:>15% to =<20% | 10
  Week 48:>20% reduction: number analyzed (Participants) | 239
  Week 48:>20% reduction | 11
  Week 48:>20% to <80%: number analyzed (Participants) | 239
  Week 48:>20% to <80% | 7
  Week 78:=<15% reduction: number analyzed (Participants) | 177
  Week 78:=<15% reduction | 160
  Week 78:>15% to =<20%: number analyzed (Participants) | 177
  Week 78:>15% to =<20% | 4
  Week 78:>20% reduction: number analyzed (Participants) | 177
  Week 78:>20% reduction | 13
  Week 78:>20% to <80%: number analyzed (Participants) | 177
  Week 78:>20% to <80% | 6
  Week 104:=<15% reduction: number analyzed (Participants) | 32
  Week 104:=<15% reduction | 32
  Week 104:>15% to =<20%: number analyzed (Participants) | 32
  Week 104:>15% to =<20% | 0
  Week 104:>20% reduction: number analyzed (Participants) | 32
  Week 104:>20% reduction | 0
  Week 104:>20% to <80%: number analyzed (Participants) | 32
  Week 104:>20% to <80% | 0
  Week 130:=<15% reduction: number analyzed (Participants) | 5
  Week 130:=<15% reduction | 4
  Week 130:>15% to =<20%: number analyzed (Participants) | 5
  Week 130:>15% to =<20% | 0
  Week 130:>20% reduction: number analyzed (Participants) | 5
  Week 130:>20% reduction | 1
  Week 130:>20% to <80%: number analyzed (Participants) | 5
  Week 130:>20% to <80% | 1
  Week 156:=<15% reduction: number analyzed (Participants) | 2
  Week 156:=<15% reduction | 2
  Week 156:>15% to =<20%: number analyzed (Participants) | 2
  Week 156:>15% to =<20% | 0
  Week 156:>20% reduction: number analyzed (Participants) | 2
  Week 156:>20% reduction | 0
  Week 156:>20% to <80%: number analyzed (Participants) | 2
  Week 156:>20% to <80% | 0

8. Primary Outcome: Number of Participants With Clinically Meaningful Change in Borg Dyspnea Score Considered as an AE
Description: Borg dyspnea score was a validated participant reported outcome assessing participant's perceived difficulty in breathing (dyspnea). The score ranges from 0 (nothing at all) to 10 (maximal difficulty). Higher scores indicated greater difficulty in breathing.
Time Frame: From Week 0 to Week 132 at specified time points
Population: The As-treated Population included participants who received at least one dose of mavrilimumab 100 mg Q2W.
Measure: Number; unit: Participants
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 394
Participants | 0

9. Primary Outcome: Oxygen Saturation Levels by Pulse Oximetry
Description: Oxygen saturation measured by pulse oximetry which measures the concentration of oxygen in the blood.
Time Frame: From Week 0 to Week 132 at specified time points
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Percent saturation
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
Percent saturation
  Week 0 (n=397) | 97.6 (0.1)
  Week 12 (n=384): number analyzed (Participants) | 384
  Week 12 (n=384) | 97.6 (0.1)
  Week 24 (n=1): number analyzed (Participants) | 1
  Week 24 (n=1) | 98.0 (NA) — Standard error was not calculated due to limited sample size.
  Week 36 (n=357): number analyzed (Participants) | 357
  Week 36 (n=357) | 97.5 (0.1)
  Week 48 (n=327): number analyzed (Participants) | 327
  Week 48 (n=327) | 97.8 (0.1)
  Week 60 (n=281): number analyzed (Participants) | 281
  Week 60 (n=281) | 97.8 (0.1)
  Week 72 (n=233): number analyzed (Participants) | 233
  Week 72 (n=233) | 97.7 (0.1)
  Week 84 (n=222): number analyzed (Participants) | 222
  Week 84 (n=222) | 97.7 (0.1)
  Week 96 (n=188): number analyzed (Participants) | 188
  Week 96 (n=188) | 97.9 (0.1)
  Week 108 (n=58): number analyzed (Participants) | 58
  Week 108 (n=58) | 97.8 (0.2)
  Week 120 (n=18): number analyzed (Participants) | 18
  Week 120 (n=18) | 97.6 (0.3)
  Week 132 (n=7): number analyzed (Participants) | 7
  Week 132 (n=7) | 97.9 (0.5)

10. Primary Outcome: Diffusing Capacity of the Lung for Carbon Monoxide (DLCO)
Description: DLCO is a pulmonary function testing that measures partial pressure difference between inspired and expired carbon monoxide.
Time Frame: From Week 12 to Week 156 at specified time points
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: (mL/min/mmHg)
Arm/Group | Mavrilimumab 100 mg
Number analyzed (Participants) | 397
(mL/min/mmHg)
  Week 12 (n=80): number analyzed (Participants) | 80
  Week 12 (n=80) | 21.196 (5.158)
  Week 24 (n=155): number analyzed (Participants) | 155
  Week 24 (n=155) | 21.996 (5.274)
  Week 48 (n=203): number analyzed (Participants) | 203
  Week 48 (n=203) | 21.135 (4.873)
  Week 78 (n=165): number analyzed (Participants) | 165
  Week 78 (n=165) | 20.639 (4.637)
  Week 104 (n=144): number analyzed (Participants) | 144
  Week 104 (n=144) | 20.636 (5.088)
  Week 130 (n=52): number analyzed (Participants) | 52
  Week 130 (n=52) | 20.372 (4.546)
  Week 156 (n=6): number analyzed (Participants) | 6
  Week 156 (n=6) | 19.265 (4.131)

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to 12 weeks after the last dose of study drug (approximately up to 3 years)
Arm/Group | Mavrilimumab 100 mg
Serious Adverse Events (participants affected / at risk) | 46/397
Other Adverse Events (participants affected / at risk) | 214/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mavrilimumab 100 mg (N=397)
Anaemia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Appendiceal abscess (Infections and infestations) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Peritonitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 2 (2)
Pyomyositis (Infections and infestations) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Myelitis transverse (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (2)
Subclavian artery thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mavrilimumab 100 mg (N=397)
Dental caries (Gastrointestinal disorders) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 15 (15)
Bronchitis (Infections and infestations) | 44 (59)
Gastroenteritis (Infections and infestations) | 11 (14)
Influenza (Infections and infestations) | 23 (26)
Nasopharyngitis (Infections and infestations) | 59 (90)
Oral herpes (Infections and infestations) | 11 (13)
Pharyngitis (Infections and infestations) | 18 (20)
Respiratory tract infection (Infections and infestations) | 13 (21)
Rhinitis (Infections and infestations) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 31 (43)
Urinary tract infection (Infections and infestations) | 35 (53)
Viral infection (Infections and infestations) | 8 (10)
Fall (Injury, poisoning and procedural complications) | 8 (8)
Alanine aminotransferase increased (Investigations) | 8 (8)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 12 (13)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 38 (78)
Headache (Nervous system disorders) | 17 (35)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Hypertension (Vascular disorders) | 26 (27)

LIMITATIONS AND CAVEATS:
The study was terminated after approximately 3 years due to future clinical development plans, including ethical considerations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.